CLINICAL TRIAL: NCT03025412
Title: A Comparison of Endoscopic Surgery and Conservative Treatment in Patients With Longstanding Mid-portion Achilles Tendinopathy
Brief Title: A Comparison of Endoscopic Surgery and Exercise Therapy in Patients With Longstanding Achilles Tendinopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties due to recently introduced new surgical procedure
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/1931
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Tendinopathy
Keywords: Achilles Tendon; Endoscopy; Minimally Invasive Surgical Procedures; Exercise therapy
MeSH Terms: conditions — Tendinopathy | interventions — Endoscopy; Physical Therapy Modalities; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic surgery (Experimental): Ambulatory surgery. Postoperative rehabilitation. From week 6 postoperative the patients start the same exercise regimen as the conservative treatment group.
  Interventions: Procedure: endoscopic surgery; Behavioral: physiotherapy and exercise
- Conservative treatment (Active Comparator): Physiotherapy and exercise. First physiotherapy consultation: Information, advice, instructions. Exercise regime during 12 weeks in three phases.
  Interventions: Behavioral: physiotherapy and exercise

INTERVENTIONS:
Procedure: endoscopic surgery — Ambulatory surgery. Same surgeon for all patients. General anesthesia. Full debridement of the paratenon and crural fascia. Also the plantaris longus tendon is debrided, but no additional tenotomy executed. Postoperative rehabilitation. Oral nonsteroidal anti-inflammatory drugs 7 days postoperatively. Active ankle dorsiflexion and plantar flexion from day 1 postoperative. Partly weight bearing (30 kg) from day 1 postoperative. Full weight bearing allowed from week 3 postoperative. Gradually increased load, both in activity of daily living, stationary bike and stretching, with individually and pragmatic progression due to pain response. From week 6 postoperative the patients start the same exercise regimen as the conservative treatment group.
  Arms: Endoscopic surgery
Behavioral: physiotherapy and exercise — Exercise schedule: Weeks 1-6, Eccentric unilateral loading while standing on the step of a staircase performed in two exercises; with straight knee and with bent knee. Weeks 7-9, Eccentric - Concentric loading while standing on the step of a staircase performed with straight knee and bent knee. Dose: 15 repetitions x 3 performed with straight knee, and 15 repetitions x 3 performed with bent knee. 3 - 4 times a week. Weeks 10-12, Eccentric - Concentric loading while standing on the step of a staircase performed with straight knee and bent knee. Dose: 15 repetitions maximum (15RM) x 3 performed with straight knee, and 15 RM x 3 performed with bent knee. 3 - 4 times a week. One leg performance or hand hold weight for extra load is used to obtain the exact number of RM.

SUMMARY:
Exercise is a preferred treatment modality for mid-portion achilles tendinopathy. Despite this, as many as 44 % of achilles tendinopathy patients do not respond to exercise treatment.

Surgery for midportion achilles tendinopathy has for many years been done as an open procedure. New knowledge resulted in a variety of minimally invasive procedures and the development of endoscopic surgery.

In this study, the effect of non-open surgery and conservative treatment (physiotherapy and exercises) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mid-portion achilles tendinopathy
* pain during at least 3 months
* decreased function (a score less than 80 on VISA-A)

Exclusion Criteria:

* Physiotherapy during previous three months
* history of major achilles trauma
* cardiovascular, respiratory, systemic, or metabolic conditions limiting exercise tolerance

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
pain using The Victorian Institute of Sports Assessment - Achilles | 3 months (immediately following 12 week exercising)
pain using The Victorian Institute of Sports Assessment - Achilles questionnaire (VISA-A) | 6 months after 12 week exercising

SECONDARY OUTCOMES:
pain using a numeric rating scale (NRS) | 3 months (immediately following 12 week exercising
pain using a numeric rating scale (NRS) | 6 months after 12 week exercising
Hospital Anxiety and Depression Scale (HAD) | 3 months (immediately following 12 week exercising)
Hospital Anxiety and Depression Scale (HAD) | 6 months after 12 week exercising
Tampa Scale of Kinesiophobia [TSK] | 3 months (immediately following 12 week exercising)
Tampa Scale of Kinesiophobia [TSK] | 6 months after 12 week exercising
Patient-clinician therapeutic relationship | 3 months (immediately following 12 week exercising)
  assessed by Scale To Assess Therapeutic Relationships in Community Mental Health Care (STAR)
Patient-clinician therapeutic relationship | 6 months after 12 week exercising
  assessed by Scale To Assess Therapeutic Relationships in Community Mental Health Care (STAR)
Maximal strength (one repetition maximum, 1RM) | 3 months (immediately following 12 week exercising)
  Measures of maximal strength will be conducted in the following manner; participants do a warm up routine where they perform 8-15 repetitions with a comfortable load. This is performed in a leg-press machine. The load is gradually increased, and the participant performs the exercise once per attempt. 3 minutes break are given in between each attempt. The heaviest load the participants manages to lift is their 1RM, and is planned to be achieved within 3-6 attempts.
Maximal strength (one repetition maximum, 1RM) | 6 months after 12 week exercising
  Measures of maximal strength will be conducted in the following manner; participants do a warm up routine where they perform 8-15 repetitions with a comfortable load. This is performed in a leg-press machine. The load is gradually increased, and the participant performs the exercise once per attempt. 3 minutes break are given in between each attempt. The heaviest load the participants manages to lift is their 1RM, and is planned to be achieved within 3-6 attempts.
Time-to-exhaustion | 3 months (immediately following 12 week exercising)
  A time-to-exhaustion test will be performed by the participants, with the same movement as described for the 1RM-test. If there is bilateral pain, the most painful side will be tested. The plantar flexion movement will be performed with a frequency of 0.5 Hz, starting with a load of 5 kg. Each minute additional 5 kg will be added until exhaustion is achieved or pain exceeds 5 on a VAS-scale. This is a common test in studies where one wish to assess aerobic endurance capacity.
Time-to-exhaustion | 6 months after 12 week exercising
  A time-to-exhaustion test will be performed by the participants, with the same movement as described for the 1RM-test. If there is bilateral pain, the most painful side will be tested. The plantar flexion movement will be performed with a frequency of 0.5 Hz, starting with a load of 5 kg. Each minute additional 5 kg will be added until exhaustion is achieved or pain exceeds 5 on a VAS-scale. This is a common test in studies where one wish to assess aerobic endurance capacity.
Physical activity level | 6 months follow-up after rehabilitation
  measured by accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Helbostad, prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Neuromedicine and Movement Science, Faculty of Medicine and Health Sciences, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided